CLINICAL TRIAL: NCT01798225
Title: The Relationships Between Periodontal Disease and Type 2 Diabetes Mellitus in the Gullah Population and the Effects of Mechanical Periodontal Therapy and Systemic Antibiotics on the Glycemic Control
Brief Title: Relationship of Periodontal Disease Treatment and Type 2 Diabetes Mellitus in the Gullah Population
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P20RR017696-06 (NIH); P20RR017696 (NIH)
Record Dates: First submitted 2012-04-18; First posted 2013-02-25 (Estimated); Results first posted 2018-10-04 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Periodontal Disease; Type 2 Diabetes Mellitus
Keywords: Periodontal Disease; Type 2 Diabetes Mellitus; Gullah African Americans
MeSH Terms: conditions — Periodontal Diseases; Diabetes Mellitus, Type 2 | interventions — Control Groups; Doxycycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): Participants received mechanical periodontal therapy, oral hygiene instructions and placebo (antibiotic) pills.
  Interventions: Drug: Placebo
- Doxycycline (Experimental): Participants received mechanical periodontal therapy, oral hygiene instructions and antibiotic (Doxycycline 100mg x 14 pills)
  Interventions: Drug: Doxycycline

INTERVENTIONS:
Drug: Placebo — Participants received mechanical periodontal therapy, oral hygiene instructions and placebo pills.
  Other Names: Control Group
  Arms: Control
Drug: Doxycycline — Participants received mechanical periodontal therapy, oral hygiene instructions and Doxycycline 100mg x 14 pills (to be taken one a day for 14 days)
  Other Names: Intervention Group
  Arms: Doxycycline

SUMMARY:
Our overall hypothesis is that treatment of periodontal disease will produce better diabetes glycemic control (glycated hemoglobin A1c, or HbA1c) and reduced levels of the catalytically active form of matrix metalloproteinase (aMMP-8) in the Gullah African American type 2 diabetes patients living on the Sea Islands of the South Carolina coast. The gingival crevicular fluid (GCF) aMMP-8 levels will be measured through a site-specific, novel noninvasive technique allowing the pathophysiological status of the periodontium tissue to be monitored. The investigators will conduct an interventional study on this population with minimal genetic admixture.

DETAILED DESCRIPTION:
Specific Aim 1: To ascertain the rate of periodontal disease progression on poorly controlled Type 2 diabetic Gullah African American patients as compared to well-controlled Gullah African American patients. The host inflammatory response appears to be the critical determinant for susceptibility and severity of marginal periodontitis especially in systemically compromised individuals13, with diabetic status perhaps increasing host susceptibility to periodontal infection due to impaired immune response14. Patients have been evaluated 6 months to one year prior to periodontal therapy (this evaluation is connected to a previous COBRE project entitled "Epidemiological Study of Periodontal Disease and Diabetes" by Dr. J. Fernandes). A reevaluation will be made at the time of periodontal therapy. Clinical periodontal parameters and HbA1c levels will be compared.

Specific Aim 2: To assess the effects of successful periodontal therapy on the level of glycemic control in this Gullah African American population. Authors addressing whether the treatment of periodontitis or other infections of the oral cavity can improve glycemic control in diabetic patients report contradictory results. We will treat periodontal patients with mechanical therapy (scaling and root planning) and oral hygiene instruction, with or without systemic antibiotic administration (Table 1). The HbA1c, fasting glucose and clinical periodontal parameters will be evaluated prior to the periodontal intervention, and at 3 and 6 months after therapy. We plan to continue to recruit, enroll and assess new patients from the Gullah African American community living on the Sea Islands of the South Carolina coast for future research projects

Specific Aim 3: To assess the concentration of the catalytically active form of MMP-8 at baseline (prior to periodontal intervention) and at 3 and 6 months later. Polymorphonuclear (PMN) leukocyte-derived MMP-8 is predominantly present in periodontitis-affected GCF9,15-16. Analysis of GCF for aMMP-8 could provide a novel useful noninvasive technique to assess and monitor the pathophysiological status of the periodontium tissue in a site-specific manner9-10.

ELIGIBILITY:
Inclusion Criteria:

* Gullah African Americans;
* With type 2 diabetes mellitus defined according to the American Diabetes Association criteria;

Other inclusion criteria are presented under each Specific Aim:

* AIM 1: Participants who have received oral, dental, periodontal, diabetes and genotype assessment through enrollment in Dr. J. Fernandes' COBRE project.
* AIM 2 and 3: Participants with severe chronic periodontitis, as defined by at least one tooth surface with probing depth (PD)≥5mm.

Exclusion Criteria:

* Severe concurrent illnesses / conditions that would limit their daily life or require extensive systemic treatment, such as malignancy, severe cardiovascular disease, organ transplant, or inadequate understanding due to mental disorders;
* Finger stick blood glucose measurement of more than 350mg/dl or less than 70mg/dl after second measurement;
* Systolic blood pressure of more than 180mm Hg or diastolic pressure of more than 100mm Hg;
* Fasting serum C-peptide < 1ng/ml (documentation or test);
* Serum creatinine ≥ 1.6mg/dl;
* Abnormal hepatic function;
* Hemoglobinopathy (sickle cell trait/hemolytic anemia) interfering with HbA1c monitoring;
* Other underlying illness/conditions which, in the doctor's judgment, may prevent patient from adherence to the study protocol;
* Unwillingness to sign the informed consent form or enter the study;
* Pregnant women;
* Patients in need of antibiotic prophylaxis prior to dental procedures or patients that have been treated with any kind of antibiotics in the past 3 months.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2007-12; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renata S. Leite, Study Director — Medical University of South Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period from 12/18/2007 to 01/12/2010. Recruitment happened from previous studies and community events.
Period: Overall Study
Arm/Group | Control | Doxycycline
Started | 57 | 56
Completed | 57 | 53
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Doxycycline | Total
Number analyzed (Participants) | 57 | 56 | 113
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 43 | 88
  >=65 years | 12 | 13 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 38 | 85
  Male | 10 | 18 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 57 | 56 | 113
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 57 | 56 | 113
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 57 | 56 | 113

OUTCOME MEASURES:

1. Primary Outcome: Glycated Hemoglobin A1c
Description: Glycated Hemoglobin A1c
Time Frame: Change between baseline to 6-month post-treatment
Measure: Mean (Full Range); unit: percentage of Glycated Hemoglobin A1c
Arm/Group | Control | Doxycycline
Number analyzed (Participants) | 57 | 56
percentage of Glycated Hemoglobin A1c | 8 [5.3 to 12.8] | 8.2 [4.7 to 14.1]

2. Primary Outcome: Periodontal Pocket Probing Depth (PD)
Time Frame: Change between baseline to 6-month post-treatment
Measure: Mean (Standard Error); unit: mm
Arm/Group | Control | Doxycycline
Number analyzed (Participants) | 57 | 56
mm | -1.98 (0.0001) | -1.37 (0.0001)

ADVERSE EVENTS:
Arm/Group | Control | Doxycycline
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/56
Other Adverse Events (participants affected / at risk) | 0/57 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No